CLINICAL TRIAL: NCT05499884
Title: Feasibility and Potential Aids of Intra-operative Endo-vaginal Ultrasound When Performing Rectal Shaving for Endometriosis
Acronym: ECHOENDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021_0273; 2022-A01264-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-08-09; First posted 2022-08-12 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Endometriosis
Keywords: deep pelvic endometriosis; rectal shaving segmental digestive resection; endovaginal ultrasound
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Procedure: Endovaginal ultrasound

INTERVENTIONS:
Procedure: Endovaginal ultrasound — Endovaginal ultrasound will be performed in the operating room by the radiology team to:
  1. to confirm the operative indication for a rectal shaving ;
  2. to confirm the complete removal of the lesion

SUMMARY:
The protocol of this study consists in the inclusion of patients with endometriosic rectal involvement with a scheduled intervention. An endovaginal ultrasound will be performed in the operating room by the radiology team to confirm the operative indication of rectal shaving then in a second step a second ultrasound in the operating room will confirm the complete excision of the lesion or the case will allow to perform a more complete gesture (discoid or segmental resection) if the shaving is not sufficient with ultrasound and / or macroscopically

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Deep pelvic endometriosis with symptomatic rectal involvement
* With surgical indication of rectal shaving validated in "RCP" or during the pre-operative consultation by the surgeon

Exclusion Criteria:

* History of inflammatory digestive pathology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with scheduled surgery for pelvic endometriosis with rectal involvement
Enrollment: 10 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Questioning the choice of surgical technique (performing a more complete procedure, such as discoid or segmental resection, immediately or after shaving) | during the procedure/surgery
  if endovaginal ultrasound performed in the operating room (before or after shaving) modifies the choice of surgical technique in at least 2 cases out of 10, the value of endovaginal ultrasound in the operating room in the management of rectal damage by shaving will be validated

SECONDARY OUTCOMES:
anatomo-pathological analysis of the operating piece. | during the procedure/surgery
  The anatomo-pathological data will be available if the choice of surgical technique is modified following one of the endovaginal ultrasound scans carried out in the operating theatre - and therefore if a discoid or segmental resection is carried out. By confirming damage to the rectal mucosa and/or stenosis of the digestive lumen, these anatomo-pathological analyses will make it possible to validate the questioning of the choice of surgical technique.
  This information is thus complementary to the main evaluation criterion, by providing an external validity criterion.

CONTACTS AND LOCATIONS:
Overall Officials: Chrystele RUBOD, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Service DE CHIRURGIE GYNECOLOGIE CHU LILLE, Lille, France